CLINICAL TRIAL: NCT01088984
Title: An Open-Label Study of Bendamustine Hydrochloride for the Treatment of Pediatric Patients With Relapsed or Refractory Acute Leukemia
Brief Title: Study of Bendamustine Hydrochloride for the Treatment of Pediatric Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/2046; 2010-020768-40 (EudraCT Number)
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Bendamustine Hydrochloride

ARMS (1):
- Bendamustine (Experimental): Bendamustine 90 or 120 mg/m^2 administered as an intravenous (IV) infusion over 60 minutes on Days 1 and 2 of each 21-day cycle (maximum of 12 total cycles), with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine

SUMMARY:
The primary objective of phase 1 of this study is to establish the recommended phase II dose (RP2D). The primary objective of phase 2 of this study is to evaluate the safety and efficacy of bendamustine at the recommended pediatric dose for the treatment of pediatric patients with relapsed or refractory acute leukemia.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has histologically proven acute lymphocytic leukemia (ALL) or acute myeloid leukemia (AML) that has relapsed or is refractory to the last regimen, and the patient is without alternative curative therapy.
* The patient's last myelosuppression therapy ended at least 2 weeks before the first dose of study drug.
* Nonhematologic acute toxic effects of prior therapy have resolved to grade 2 or less according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
* The patient has adequate liver function with bilirubin values less than or equal to 1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) values less than or equal to 5 times the age-appropriate ULN.
* The patient has adequate renal function with serum creatinine values less than 2 times ULN.
* The patient has Karnofsky or Lansky performance status of 60 or greater. Patients older than 16 years of age will be scored according to the Karnofsky scale and patients 16 years of age or younger will be scored according to the Lansky scale.
* The patient may have had hematopoietic stem cell transplantation.
* Women of childbearing potential (not surgically sterile) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of treatment and for 30 days after the end of treatment.
* Men not surgically sterile or who are capable of producing offspring must practice abstinence or use a barrier method of birth control, and must agree to continue use of this method for the duration of treatment and for 30 days after the end of treatment.
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Key Exclusion Criteria:

* The patient has any active, uncontrolled systemic infection, severe concurrent disease, or symptomatic untreated central nervous system (CNS) involvement.
* The patient has evidence of active graft versus host disease.
* The patient has a known human immunodeficiency virus (HIV) infection.
* The patient has active hepatitis B or hepatitis C infection.
* The patient is a pregnant or lactating woman. Any women becoming pregnant during the study will be withdrawn from the study immediately.
* The patient has any serious uncontrolled medical or psychological disorder that would impair the ability of the patient to receive study drug.
* The patient has any condition that places the patient at unacceptable risk or confounds the ability of the investigators to interpret study data.
* The patient has received any other investigational agent within 30 days of study entry.
* The patient has known hypersensitivity to bendamustine or mannitol.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (50):
- United States (19):
  - Teva Investigational Site 17, Orange, California
  - Teva Investigational Site 12, San Diego, California
  - Teva Investigational Site 10, St. Petersburg, Florida
  - Teva Investigational Site 8, Baltimore, Maryland
  - Teva Investigational Site 16, Boston, Massachusetts
  - Teva Investigational Site 9, Detroit, Michigan
  - Teva Investigational Site 1, Jackson, Mississippi
  - Teva Investigational Site 5, Kansas City, Missouri
  - Teva Investigational Site 14, St Louis, Missouri
  - Teva Investigational Site 15, New York, New York
  - Teva Investigational Site 18, Portland, Oregon
  - Teva Investigational Site 11, Hershey, Pennsylvania
  - Teva Investigational Site 7, Philadelphia, Pennsylvania
  - Teva Investigational Site 19, Memphis, Tennessee
  - Teva Investigational Site 3, Dallas, Texas
  - Teva Investigational Site 4, Fort Worth, Texas
  - Teva Investigational Site 13, Houston, Texas
  - Teva Investigational Site 2, Seattle, Washington
  - Teva Investigational Site 6, Milwaukee, Wisconsin
- Australia (3):
  - Teva Investigational Site 300, Herston
  - Teva Investigational Site 301, Parkville
  - Teva Investigational Site 302, Randwick
- Teva Investigational Site 520, Minsk, Belarus
- Brazil (8):
  - Teva Investigational Site 615, Barretos-SP
  - Teva Investigational Site 616, Caxias do Sul
  - Teva Investigational Site 613, Curitiba-PR
  - Teva Investigational Site 612, Porto Alegre
  - Teva Investigational Site 614, Porto Alegre
  - Teva Investigational Site 617, Sao Paulo-SP
  - Teva Investigational Site 610, São Paulo
  - Teva Investigational Site 611, São Paulo
- Teva Investigational Site 100, Toronto, Canada
- Israel (3):
  - Teva Investigational Site 501, Jerusalem
  - Teva Investigational Site 503, Petah Tikva
  - Teva Investigational Site 502, Ramat Gan
- Mexico (4):
  - Teva Investigational Site 603, Guadalajara
  - Teva Investigational Site 600, Mexico City
  - Teva Investigational Site 601, Mexico City
  - Teva Investigational Site 602, Monterrey
- Teva Investigational Site 303, Auckland, New Zealand
- Poland (3):
  - Teva Investigational Site 531, Bialystok
  - Teva Investigational Site 530, Lublin
  - Teva Investigational Site 532, Warsaw
- Russia (2):
  - Teva Investigational Site 511, Moscow
  - Teva Investigational Site 510, Saint Petersburg
- Teva Investigational Site 320, Singapore, Singapore
- South Korea (4):
  - Teva Investigational Site 330, Seoul
  - Teva Investigational Site 331, Seoul
  - Teva Investigational Site 332, Seoul
  - Teva Investigational Site 333, Seoul

REFERENCES:
- [Background] Fraser C, Brown P, Megason G, Ahn HS, Cho B, Kirov I, Frankel L, Aplenc R, Bensen-Kennedy D, Munteanu M, Weaver J, Harker-Murray P. Open-label bendamustine monotherapy for pediatric patients with relapsed or refractory acute leukemia: efficacy and tolerability. J Pediatr Hematol Oncol. 2014 May;36(4):e212-8. doi: 10.1097/MPH.0000000000000021. PMID 24072240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 46 patients screened, 43 patients at 24 centers from the United States, Australia, South Korea, Israel, Mexico, and Brazil met entry criteria and were considered eligible for enrollment. Of the 3 patients who were not enrolled, 2 patients died prior to study enrollment, and 1 patient was ineligible because inclusion criteria were not met.
Groups:
- Bendamustine 90 mg/m^2: Bendamustine 90 mg/m^2 administered as an intravenous (IV) infusion over 60 minutes on Days 1 and 2 of a 21-day Induction cycle, with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
- Bendamustine 120 mg/m^2: Bendamustine 120 mg/m^2 administered as an IV infusion over 60 minutes on Days 1 and 2 of each 21-day cycle (maximum of 12 total cycles), with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
Period: Phase 1
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Started | 5 | 6
Completed | 0 (completed follow-up up to 12 month from last dose of study drug) | 0 (completed follow-up up to 12 month from last dose of study drug)
Not Completed | 5 | 6
Not completed — Death | 2 | 1
Not completed — Disease Progression | 2 | 4
Not completed — Other | 1 | 1
Period: Phase 2
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Started | 0 | 32
Completed | 0 (completed follow-up up to 12 month from last dose of study drug) | 0 (completed follow-up up to 12 month from last dose of study drug)
Not Completed | 0 | 32
Not completed — Death | 0 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — DIsease Progression | 0 | 25
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes 5 participants treated with bendamustine at 90 mg/m2 in Phase 1, and 6 participants treated with bendamustine at 120 mg/m2 in Phase 1, and 32 participants treated with the recommended phase II dose (RP2D) of bendamustine (120 mg/m2) in Phase 2.
Groups:
- Phase 1: Bendamustine 90 or 120 mg/m^2: Bendamustine 90 or 120 mg/m^2 administered as an IV infusion over 60 minutes on Days 1 and 2 of a 21-day Induction Cycle, with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
- Phase 2: Bendamustine 120 mg/m^2: Bendamustine 120 mg/m^2 administered as an IV infusion over 60 minutes on Days 1 and 2 of each 21-day cycle (Cycles 2 through 12), with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Bendamustine 90 or 120 mg/m^2 | Phase 2: Bendamustine 120 mg/m^2 | Total
Number analyzed (Participants) | 11 | 32 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.31) | 9.3 (4.93) | 9.2 (4.74)
Age, Customized [Number; unit: participants]
  1 to 6 years | 4 | 10 | 14
  7 to 11 years | 3 | 10 | 13
  12 to 20 years | 4 | 12 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 12 | 13
  Male | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D) of Bendamustine
Description: RP2D was determined by a traditional 3+3 dose escalation design, with the following restrictions: only doses of 60, 90, 120, and 150 mg/m^2 were explored, and escalation to 150 mg/m^2 would only occur if the 120 mg/m^2 dose was deemed safe and pharmacokinetic data indicate subtherapeutic exposure as compared with adults. The first cohort was administered bendamustine at the 90 mg/m^2 dose; de-escalation to the 60 mg/m^2 dose would only occur if the starting dose led to dose-limiting toxicity (DLT) in 2 or more participants. A DLT was defined as any study drug-related nonhematologic adverse event (AE) that was grade 4 for toxicity by National Cancer Institute's Common Toxicity Criteria for AEs, version 4. In addition, grade 3 or above allergic reaction or skin rash were considered DLTs. Hematologic AEs were not considered DLTs. The dose level at which at least 2 of 3 or 2 of 6 participants had a DLT was considered as exceeding the RP2D. The RP2D was the dose 1 step below that level.
Time Frame: Induction Cycle (21- to 35-day cycle)
Population: All participants enrolled in Phase 1 of the study.
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1: Bendamustine 90 or 120 mg/m^2
Number analyzed (Participants) | 11
mg/m^2 | 120

2. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was calculated as follows: number of participants in the primary analysis set achieving a best overall response of complete remission without platelet recovery (CRp) or complete remission (CR), divided by the number of participants in the primary analysis set. The most positive response for each patient during the study was counted. The 95% CI was calculated using binomial parameter exact method. Response was determined by the investigator, and evaluated per Jeha et al, 2006: A CR required no evidence of circulating blasts or extramedullary disease, an M1 marrow (≤ 5% bone marrow blasts), and recovery of peripheral counts (platelets ≥ 100 × 10^9/L and absolute neutrophil count ≥ 1.0 × 10^9/L). A CR without platelet recovery (CRp) required all of the criteria for a CR with the exception of platelet recovery.
Time Frame: Assessed at each treatment cycle (21 to 35 days), for a maximum of 12 cycles
Population: The primary analysis set for efficacy included all participants treated at the RP2D in Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Bendamustine 120 mg/m^2
Number analyzed (Participants) | 32
percentage of participants | 0 [0.00 to NA] — 1-sided 95% confidence interval
Statistical Analysis 1: Comparison: Phase 2: Bendamustine 120 mg/m^2; Test type: Superiority or Other; p = 1.0000, binomial parameter exact method — 1-sided p-value is calculated against the null hypothesis of a response rate of 5%

3. Secondary Outcome: Best Overall Tumor Response Rate
Description: Biological activity of bendamustine was defined as achieving a best response of partial response (PR), CRp, or CR. Rate was calculated as follows: number of participants in the primary analysis set achieving a best overall response of PR, CRp, or CR, divided by the number of participants in the primary analysis set. The most positive response for each patient during the study was counted. The 95% CI was calculated using binomial parameter exact method. Response was determined by the investigator, and evaluated per Jeha et al, 2006: A PR had to meet the following criteria: complete disappearance of circulating blasts and an M2 marrow (≥ 5% and ≤ 25% bone marrow blasts) and appearance of normal progenitor cells or an M1 marrow that did not qualify for CR or CRp. See Outcome Measure 2 for full definitions for CRp and CR.
Time Frame: At each treatment cycle (21 to 35 days), for a maximum of 12 cycles
Population: The primary analysis set for efficacy included all participants treated at the RP2D in Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Bendamustine 120 mg/m^2
Number analyzed (Participants) | 32
percentage of participants | 6 [0.77 to 20.81]

4. Secondary Outcome: Best Overall Tumor Response Rate, by Phase
Description: as for outcome 3
Time Frame: At each treatment cycle (21 to 35 days), for a maximum of 12 cycles
Population: The safety analysis set included all participants treated at any dose of bendamustine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: Bendamustine 90 or 120 mg/m^2 administered as an IV infusion over 60 minutes on Days 1 and 2 of each 21-day cycle (maximum of 12 total cycles), with delays up to 2 weeks for neutrophil and platelet count recovery, for up to a 35-day cycle.
Arm/Group | Phase 1: Bendamustine 90 or 120 mg/m^2 | Phase 2: Bendamustine 120 mg/m^2 | Total
Number analyzed (Participants) | 11 | 32 | 43
percentage of participants | 18 [2.28 to 51.78] | 6 [0.77 to 20.81] | 9 [2.59 to 22.14]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was determined for the participants with CR or CRp in the primary analysis set, defined as the time from first achieving remission to the time when progression was diagnosed, the participant died, or the participant started receiving new antineoplastic therapy. Data from participants who do not progress were censored at the last valid assessments. Median DOR and its 95% confidence interval was determined based on the Kaplan-Meier method. Data from participants who received a transplant were censored at the time of the transplant.
Time Frame: At each treatment cycle (21 to 35 days), for a maximum of 12 cycles
Population: No duration of remission (defined as CR or CRp) analysis was performed for participants in the primary analysis since none achieved remission.
Arm/Group | Phase 2: Bendamustine 120 mg/m^2
Number analyzed (Participants) | 0

6. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) for Bendamustine and Its Metabolites (M3 and M4)
Time Frame: Cycle 1, Day 1: before infusion, immediately following the infusion, and 3, 6, 10(±2), and 24 hours after the start of infusion. The 24-hour postinfusion sample was obtained before the start of the infusion on Day 2.
Population: The pharmacokinetic analysis set included all participants who were in the safety analysis set (ie, those treated at any dose of bendamustine) who had valid pharmacokinetic data; n=number of participants with valid data for this assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Number analyzed (Participants) | 5 | 37
ng/mL
  Bendamustine; n=5, 37 | 5093.24 (60.39) | 6401.80 (52.90)
  Metabolite M3; n=5, 36 | 311.70 (92.98) | 403.52 (69.91)
  Metabolite M4; n=5, 37 | 37.53 (82.97) | 48.27 (53.94)

7. Secondary Outcome: Time to Maximum Plasma Drug Concentration (Tmax) for Bendamustine and Its Metabolites (M3 and M4)
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Number analyzed (Participants) | 5 | 37
hours
  Bendamustine; n=5, 37 | 1.14 (10.00) | 1.07 (9.49)
  Metabolite M3; n=5, 36 | 1.14 (10.00) | 1.07 (9.53)
  Metabolite M4; n=5, 37 | 1.14 (10.00) | 1.07 (9.49)

8. Secondary Outcome: Area Under the Plasma Drug Concentration by Time Curve From Time 0 Until the Last Measurable Plasma Concentration (AUC0-t) for Bendamustine and Its Metabolites (M3 and M4)
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Number analyzed (Participants) | 5 | 37
ng*hr/mL
  Bendamustine; n=5, 37 | 11174.86 (51.73) | 11046.32 (58.58)
  Metabolite M3; n=5, 36 | 697.09 (88.37) | 701.19 (67.38)
  Metabolite M4; n=5, 37 | 43.80 (109.72) | 72.78 (57.11)

9. Secondary Outcome: Area Under the Plasma Drug Concentration by Time Curve From Time 0 Until 24 Hours After Study Drug Administration (AUC0-24) for Bendamustine and Its Metabolites (M3 and M4)
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Bendamustine 90 mg/m^2 | Bendamustine 120 mg/m^2
Number analyzed (Participants) | 5 | 37
ng*hr/mL
  Bendamustine; n=1, 13 | 14998.00 (NA) — only 1 participant assessed | 12929.22 (50.46)
  Metabolite M3; n=0, 2 | NA (NA) — no participants assessed | 1336.89 (1.80)
  Metabolite M4; n=0, 0 | NA (NA) — no participants assessed | NA (NA) — no participants assessed

ADVERSE EVENTS:
Time Frame: Screening (Day -14 to Day-1) through end of treatment (up to 12 35-day cycles), plus 30 days.
Description: Participants were given both dosages for varying lengths and the adverse events were not reported according to which timepoint neither at which dosage events occurred.
Arm/Group | Bendamustine
Serious Adverse Events (participants affected / at risk) | 33/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (13)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (2)
Pyrexia (General disorders) | 4 (7)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Aspergillosis (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1)
Capnocytophagia infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Febrile infection (Infections and infestations) | 1 (1)
Fungal sepsis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=43)
Anaemia (Blood and lymphatic system disorders) | 28 (92)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (19)
Lymphopenia (Blood and lymphatic system disorders) | 3 (10)
Neutropenia (Blood and lymphatic system disorders) | 5 (8)
Pancytopenia (Blood and lymphatic system disorders) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (74)
Abdominal pain (Gastrointestinal disorders) | 9 (13)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 14 (28)
Gingival bleeding (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 20 (26)
Vomiting (Gastrointestinal disorders) | 15 (31)
Catheter site pain (General disorders) | 3 (3)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 3 (3)
Fatigue (General disorders) | 7 (10)
Mucosal inflammation (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 4 (10)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 21 (35)
Bacteraemia (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 6 (11)
Blood creatinine increased (Investigations) | 5 (20)
Blood potassium decreased (Investigations) | 3 (13)
Platelet count decreased (Investigations) | 8 (41)
Weight decreased (Investigations) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 9 (12)
Fluid overload (Metabolism and nutrition disorders) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (40)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (15)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 9 (12)
Anxiety (Psychiatric disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Hypertension (Vascular disorders) | 12 (19)
Hypotension (Vascular disorders) | 8 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution must submit proposed publication to Sponsor for review within a prespecified number of days before submission for publication. If Sponsor's review shows that potentially patentable subject matter would be disclosed, publication/public disclosure shall be delayed to enable Sponsor, or Sponsor's designees, to file necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.